CLINICAL TRIAL: NCT05840679
Title: Effect of Different Concentrations of Sodium Hypochlorite on Post Operative Pain Following Single Visit Root Canal Treatment
Brief Title: Different Concentrations of Sodium Hypochlorite Affecting Post-endodontic Pain
Acronym: NaOCl
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Kanza Zafar, Dr. Kanza Zafar, Principal Investigator and Resident Operative Dentistry and Endodontics, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sodium Hypochlorite NaOCl
Record Dates: First submitted 2023-04-05; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 3% NaOCl concentration group (Experimental): Participants in this group will receive endodontic irrigation with lower conc 3% sodium hypochlorite
  Interventions: Drug: Irrigation Solution
- 6% NaOCl concentration group (Experimental): Participants in this group will receive endodontic irrigation with higher conc 6% sodium hypochlorite
  Interventions: Drug: Irrigation Solution

INTERVENTIONS:
Drug: Irrigation Solution — Different concentrations of NaOCl are being used as the endodontic irrigant.
  Other Names: Root Canal Disinfection

SUMMARY:
This is a randomized, prospective, double-blind, clinical trial to assess the effect of 3% and 6% sodium hypochlorite (NaOCl) as irrigant on postendodontic pain and rescue medication intake following single visit root canal treatment

DETAILED DESCRIPTION:
Diagnostic procedures to include history taking and clinical and radiographic examination with all findings being recorded in patient's notes.

• A prolonged exaggerated response (more than 10 seconds) to a cold pulp sensibility test and a positive response to the electric pulp tester will be considered evidence for irreversible pulpitis.

Patients will be asked to rate their pre-treatment pain on a visual analogue scale from 0 to 10.

Patients with moderate pain will be selected, VAS score (4 - 6).

* ANESTHESIA Patients receive 2 cartridges of 2% Articaine with 1:80000 epinephrine in an Inferior Alveolar Nerve Block Injection
* Access opening, isolation and first rinse with NaOCl After access preparation, each tooth will be isolated using rubber dam. Patients will be randomly assigned to either of the following groups: 3% NaOCl or 6% NaOCl. The pulp chamber will be filled with 2mL irrigant for 2 min followed by saline irrigation.
* Hand Instrumentation The patency of canals will be established and an initial glidepath be prepared using size 10 and 15 K-files (Mani, Mani Inc., Tochigi, Japan)
* WORKING LENGHT WL will be determined using apex locator (DentaPort ZX, J.Morita USA) and confirmed radiographically to be 1 mm short of the radiographic apex.
* ROTARY INSTRUMENTATION Mechanical prep using a Niti rotary system (Protaper Universal, Dentsply Sirona) in a torque-controlled endodontic motor (X-Smart plus, Dentsply Maillefer) according to the manufacturer's sequence and recommendations of speed and torque. Canal prep with S1 and SX instruments in a crown-down sequence to shape the coronal two-thirds of canal.
* APICAL PREPARATION Apical patency will be maintained with a size 10 K file before each rotary-instrument change.The apical preparation will be done using S1, S2, F1 or F2 up to WL corresponding to tip size of F1 or F2.
* IRRIGATION
* Between instruments, the root canals will be irrigated with 2 mL of either 3% or 6% NaOCl with a 30G x 25mm side-perforated needle (Medic Endo Irrigation Needles, HDS).
* The tip of the needle will be kept 4mm short of WL. The needle will be repeatedly moved up and down in order to prevent locking in the canals.
* Volume of irrigant use after every instrumentation - 2ml
* Total volume of NaOCl used per canal - 8-10ml , per Tooth - 24 - 30 ml
* After NaOCl, canals will be flushed with 5ml normal saline irrigation.
* Smear layer will be removed by irrigation with 17% EDTA, (EDTA; Glycle File Prep, Dentsply Maillefer) followed by 5 mL normal saline irrigation.
* DRYING CANALS At the same visit, the root canals will be dried with paper points (GAPADENT Absorbent paper points)
* OBTURATION Shall be filled with matched size gutta-percha cones (Meta Biomed Co, Korea) and sealar (Endoplus Root Canal Sealer 13,5g President Dental Germany) using the single cone technique.
* Sealed with Temporary restoration (Cavit, 3M ESPE, Germany) Patients will receive a rescue bag of 10 Ibuprofen in case they have pain with instructions for ondemand use.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between 18 to 55 years
* First and second mandibular molar diagnosed with irreversible pulpitis due to caries
* Patients with moderate pain will be selected, VAS score (4 - 6).
* Normal periapical radiographic appearance
* Mild tender to percussion
* No allergies to articaine

Exclusion Criteria:

* Patients who have taken analgesic or anti-inflammatory drugs within 6 hours before treatment visit
* Pregnant or lactating patients
* Teeth with severe periodontal disease
* Teeth that cannot be isolated with rubber dam
* Teeth undergone over-instrumentation or overfilling beyond apex
* Teeth with calcifications/ resorptive defects
* History of allergy to any materials used in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain after root canal treatment | 1 week
  Post-operative pain will be assessed using a self-report questionnaire using a numerical visual analogue scale (VAS) from 0 to 10.
  0 = No pain
  1 - 3 = Mild pain 4 - 6 = Moderate pain 7 -10 = Severe pain Pain recording will be done after 6hrs, 12hrs, 24hrs, 48hrs and 72 hrs. (Participants to be contacted by the investigator at each time point to check on them and remind them to record their pain) The given questionnaire shall be collected when the participant comes for final restoration one week later.

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Institue Of Dentistry, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No